CLINICAL TRIAL: NCT00000397
Title: Behavioral Insomnia Therapy for Fibromyalgia Patients
Brief Title: Behavioral Insomnia Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00008633; R21AR046094 (NIH); NIAMS-039
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2005-12

CONDITIONS: Fibromyalgia; Insomnia
Keywords: Fibromyalgia; Insomnia; Cognitive-behavioral therapy (CBT); Behavioral insomnia therapy
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Behavioral: Behavioral insomnia therapy

SUMMARY:
This study tests the effectiveness of a nondrug treatment for the insomnia that often occurs in people with fibromyalgia. The treatment is a type of psychotherapy called cognitive-behavioral therapy. Cognitive-behavioral therapy combines cognitive therapy, which can modify or eliminate thought patterns contributing to the person's symptoms, and behavioral therapy, which aims to help the person change his or her behavior.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a prevalent and debilitating condition that contributes to impaired occupational and social functioning and increased disability among affected individuals. The vast majority of people with FM experience persistent sleep disturbances (e.g., onset difficulty, repeated or extended awakenings, nonrestorative sleep) that worsen other FM-related symptoms (e.g., chronic pain, fatigue) and sustain their general dysfunction. Pharmacologic treatments (e.g., antidepressants, hypnotics) may reduce symptoms for some people with FM, but many FM patients display little enduring improvement in their sleep and other FM-related symptoms in response to such agents.

Our clinical observations and initial pilot work suggest that factors common among other insomnia subtypes such as conditioned bedtime arousal, erratic sleep/wake scheduling, and spending too much time in bed likely perpetuate the sleep problems of these medication-refractory FM patients. Over the past decade, we have developed, refined, and repeatedly tested a cognitive-behavioral therapy (CBT) that has proven effective for reducing sleep disturbances perpetuated by such underlying cognitive/behavioral mechanisms. The major objectives of this project are to conduct a prospective randomized clinical trial to confirm these preliminary findings and to determine the efficacy of CBT insomnia treatment for interrupting the disturbed nocturnal sleep and daytime pain, fatigue, and distress symptom complex that defines FM.

One arm of this study's three-by-four factorial design will compare CBT with both a contact control treatment and standard care. The other arm in the design is a repeated-measures factor consisting of four time points (i.e., baseline, mid-treatment, post-treatment, and 6-month follow-up periods) at which we will assess outcome. We will assess participants at all four time points with objective (wrist actigraphy) and subjective (sleep logs, Insomnia Symptom Questionnaire) measures of sleep improvements, measures of subjective pain, and questionnaires that assess mood (State-Trait Anxiety and Beck Depression Scales) and general quality of life (SF-36). We will conduct multivariate statistical analyses and tests of clinical significance with these various measures. We will also conduct exploratory analyses to determine if polysomnographically-derived sleep measures obtained prior to treatment correlate with initial levels of pain and distress or eventual treatment outcome.

Results should provide information about the usefulness of CBT for treating FM-related sleep difficulties. Results should also improve understanding of the FM syndrome in general and provide new information about the potential role of behavioral therapy in the overall management of this disorder.

Individuals interested in participating in this study should live within reasonable commuting distance from the Duke University Medical Center (Durham, NC), because this research requires multiple outpatient visits for screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia for more than 1 month
* Fibromyalgia diagnosis
* Participants must live within easy commuting distance of Duke Medical Center, Durham, North Carolina

Exclusion Criteria:

* Terminal illness
* Major psychiatric disorder
* Substance abuse
* Dependence on hypnotic drugs
* Other sleep disorders (sleep apnea, restless legs, etc.)
* Other sleep-disturbing medical disorders (painful arthritis, thyroid condition, etc.)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 1999-07; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Edinger, PhD, Principal Investigator — VA Medical Center-Durham
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Krystal AD, Edinger J, Wohlgemuth W, Marsh GR. Sleep in peri-menopausal and post-menopausal women. Sleep Med Rev. 1998 Nov;2(4):243-53. doi: 10.1016/s1087-0792(98)90011-9. PMID 15310495
- [Result] Edinger JD, Wohlgemuth WK, Krystal AD, Rice JR. Behavioral insomnia therapy for fibromyalgia patients: a randomized clinical trial. Arch Intern Med. 2005 Nov 28;165(21):2527-35. doi: 10.1001/archinte.165.21.2527. PMID 16314551